CLINICAL TRIAL: NCT03155490
Title: Translating Simulation-based Team Leadership Training Into Patient-level Outcomes
Brief Title: Study of Team Leadership Training Effect on Patient Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Michigan State University (Other); University of Maryland (Other)
Responsible Party: Principal Investigator, Rosemarie Fernandez, MD, Associate Professor, Emergency Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000748
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Wounds and Injuries; Trauma
Keywords: Hospital medical emergency team; Leadership; Simulation training
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leadership Training (Experimental): Subjects are resident trainees with a role in the emergency department evaluation and management of trauma patients.
  Interventions: Behavioral: Leadership training
- Control (No Intervention): Subjects are resident trainees with a role in the emergency department evaluation and management of trauma patients.

INTERVENTIONS:
Behavioral: Leadership training — Subjects randomized to the experimental arm of the study will receive an additional 4 hours of simulation-based trauma team leadership training. This training is in addition to the baseline 2 hours of trauma leader training and orientation all subjects receive.
  Arms: Leadership Training

SUMMARY:
Brief Summary: Trauma is a major public health burden; it is the fifth most common cause of mortality overall in the US and accounts for the majority of deaths in patients younger than 45. Trauma resuscitations present unique patient care challenges due to the need to perform complex tasks under uncertain and time-pressured conditions. It is not entirely surprising that one-third to one-half of trauma patient-related errors occurred in emergency departments during the initial resuscitation period. Effective team leadership can enhance teamwork and team adaptability, thus improving teams' ability to handle unexpected and rapidly changing situations. Simulation-based training provides a clinically relevant practice environment that has been recommended for team and team leader training.

The purpose of this research is to evaluate the impact of simulation-based leadership training on clinical teamwork, team leadership and patient care. The investigators hypothesize that team leadership training will improve team leadership, teamwork, and critical patient care events during actual trauma resuscitations.

DETAILED DESCRIPTION:
Detailed Description: This study will implement an individual randomized controlled trial. Eligible trainee subjects (second or third year emergency medicine or general surgery residents) will be randomized within each month in a 1:1 proportion to either the intervention (team leadership training) or control (no training) conditions. Subjects will be randomized each month to ensure that outcomes are not biased by opportunities for concurrent learning throughout the residency year. The primary outcome is team leadership during actual trauma resuscitations. The secondary outcome is patient care during actual trauma resuscitations. Primary hypotheses include that the intervention group will demonstrate improved leadership (H1) and patient care (H2) during actual trauma resuscitations. The investigators will collect baseline data (pre-intervention, first 2 weeks of the month) and post-intervention/control data (last 2 weeks of the month).

Control Condition: Subjects randomized to the control condition will receive a standard orientation to the trauma team leader role at the start of their month in the ED. This orientation involves review of key administrative information, including departmental policy on chart completion, attendance policy, and available resources. No further formal trauma or team leader training will be provided for the control group.

Intervention Condition: Subjects randomized to the intervention arm of the study will also receive the standard orientation to the trauma leader role at the start of their trauma leader month in the ED. The study coordinator will then schedule these subjects for the leadership training intervention to start 11-13 days after the start of the rotation. Subjects will attend a session where they will complete the demonstration-based training and simulation-based training (simulation + debriefing + additional practice, 4 hours total) curriculum. A Laerdal SimMan 3G patient simulator and trained confederates (team members) will operationalize the resuscitation scenario. The investigators will record all simulations to allow for video-assisted debriefing and opportunity for self-reflection.

Trauma resuscitations will take place at Harborview Medical Center, an urban, tertiary care center affiliated with the University of Washington Medical Center that serves as the sole trauma center for a 5-state region (AK, WA, WY, MT, ID). Dedicated trauma resuscitation bays are equipped for all levels of trauma resuscitations. Data collection during clinical assessments will involve video recording of ongoing trauma resuscitations within two resuscitation bays. All patients presenting to the ED with a trauma-related complaint will be screened using inclusion and exclusion criteria (below). Criteria were chosen to ensure a broad representation of trauma patient care and adequate opportunity to observe team leader behaviors. Certain exclusion criteria (c-g) were selected to try to identify those patients with near 100% mortality or those inappropriate for resuscitative efforts. Additionally, pediatric and pregnant patients will be excluded as their team composition differs markedly from those involved in standard adult trauma resuscitations. Criteria will be further honed and tested prior to data collection to ensure eligible resuscitations are reliably identified and appropriate for the proposed research.

Measures Primary Outcome: Team leadership Trained raters will code video recordings of actual trauma resuscitations using a team leadership rating scale that will produce a single leadership score for each resuscitation. Raters will be blinded to study arm and will have no prior history of interaction with the subject as a physician provider. Leadership rating dimensions will be summed and averaged to create a reliable overall indicator for each trauma case. Aggregation of the multiple trauma case assessments is necessary to both create reliable indicators across trauma cases and to align the level of the data with the unit of observation and the level of analysis (i.e., the subject team leader).

Secondary Outcome: Patient care Trained raters will code video recordings of actual trauma resuscitations using a patient care rating scale that will produce a single patient care score for each resuscitation. Raters coding patient care will be distinct from those coding team leadership to minimize bias. Raters will be blinded to study arm and will have no prior history of interaction with the subject as a physician provider. Patient care rating dimensions will be summed and averaged to create a reliable overall indicator for each trauma case. Aggregation of the multiple trauma case assessments is necessary to both create reliable indicators across trauma cases and to align the level of the data with the unit of observation and the level of analysis (i.e., the subject team leader).

Patient Outcomes (Pilot) are defined below.

Analysis (Data Preparation)

Leadership and patient care rating dimensions will be summed and averaged to create a reliable overall indicator for each primary dependent variable for each trauma case. The sub-dimension ratings for each factor are on the same metric, so the combination of the rating dimensions into an overall composite indicator is straightforward.

Control composites for the subject (team leader) and patient will be examined. The investigators will first determine whether candidate control variables are associated with the primary criteria. Those candidate control variables that significantly relate to leadership behavior or patient care will be retained as controls. For retained variables, the investigators will first transform the raw control variable metrics into standardized scores to equalize their means and standard deviations. The standardized indicators will then be summed and averaged to compute control composites for the subject (team leader) and patient. Aggregation of the multiple trauma case assessments and controls (patient) is necessary to both create reliable indicators across trauma cases and to align the level of the data with the unit of observation and the level of analysis (i.e., the subject team leader). Aggregation of the patient outcome assessments will be accomplished by summing and averaging the pre- and post-interventions separately. Aggregation of the patient controls will be accomplished by summing and averaging the patient control composites.

Descriptive statistics will be used to provide univariate summaries of the basic characteristics of the team leader subjects and patients. These summaries will also be used to identify outliers and to determine if randomization resulted in the composition of study groups with similar characteristics.

Analysis (Primary and Secondary Outcomes) With the data prepared and aligned to the unit of observation, the experimental design is structured as a fixed effects two-condition pre- and post-intervention model. The analyses will contrast an intervention group receiving leadership training with a control group receiving no training, controlling for relevant subject (team leader) and patient factors and for pre-intervention subject performance. To provide a measure of control for the overall Type I experiment-wise rate the investigators will first conduct a Multivariate Analysis of Covariance (MANCOVA) that will assess the significant effect of training condition on the set of dependent variables (leadership and patient care). A significant effect at the designated alpha level (.05), will trigger follow up univariate analyses for each hypothesis (i.e., dependent variable) using Analysis of Covariance (ANCOVA).

The study was powered to address the impact of leadership training on leadership. The ability to detect significant effects in an experiment depends on the target level of statistical significance (alpha), sample size, and effect sizes of the experimental treatments. Given that our research foci are innovative, estimating anticipated effect sizes represents the major challenge for conducting a power analysis. A meta-analysis of leadership training/development programs was consulted to estimate the effect size for leadership training. Based on 35 studies with a total sample size of 3389, a mean effect size (Cohen's d, corrected for sampling error and measurement error) of .65 was found for leadership training and all outcome criteria. Using this effect size, a power analysis indicated a sample size of 60 (30 per condition) would provide .80 power in detecting true effects.

Pilot Outcome Analysis

Linkage: Assessed as the proportion of patients treated by study subjects (control and intervention groups) linked to vital status at discharge after traumatic injury. Assessed will be proportions linked to each of these groups as well as overall.

Interim Analyses: As this is a feasibility study to characterize linkage, there will be no formal interim analyses that would allow stopping the study for either efficacy or futility.

Efficacy Analyses: The linkage rate will be summarized as a binomial proportion. Secondary measures will be summarized descriptively, as recommended for pilot studies. Sample Size: A sample size of 160 eligible patients will allow estimation of linkage from simulation intervention to hospital outcome with a precision (as measured by half-width of 95% CI) of 7.7%.

ELIGIBILITY:
Inclusion Criteria:

1. Second or third year emergency medicine or general surgical resident in good standing with the Office of Graduate Medical Education
2. Up-to-date ATLS-certification
3. >6 weeks prior experience in trauma care at Harborview Medical Center
4. Scheduled for a trauma team leader month during the data collection period of the study

Exclusion Criteria:

a) Unavailable for intervention or assessment

****************************************

The trauma patients that are NOT the subjects for this study but who are the clinical recipients of subjects' care also have inclusion/exclusion criteria. These are:

Inclusion Criteria:

1. Age > 21
2. Patients with one or more of the following clinical presentations:

i. Witnessed trauma with intubation in the pre-hospital setting ii. Witnessed trauma with hypotensive (SBP< 90 mmHg for two consecutive readings) in the pre-hospital setting iii. Stab wound or impalement to the neck, chest, abdomen, pelvis, or groin iv. MVC with ejection from the vehicle v. Fall > 20ft vi. Pedestrian struck by a motorized vehicle vii. Motorcycle crash > 20 mph viii. Gunshot wounds to the head, neck, chest, abdomen, pelvis, or groin ix. Two or more obvious long bone/ extremity injuries

Exclusion Criteria:

1. Prisoners
2. Obstetric patient
3. Patient status downgraded based on first 5 min. of evaluation
4. Patient dead on arrival to ED or pronounced dead within 5 min of arrival
5. Patient removed from ED within 5 minutes of arrival
6. Patients arriving to the ED with do not resuscitate or comfort care orders
7. Patients on whom resuscitative efforts ceased within 5 minutes of arrival to the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Team leadership | Data will be collected pre- and post-intervention for approximately 5 weeks total.
  Subject performance during trauma resuscitations is video recorded and assessed using team leadership measure (behaviorally anchored rating scale). Final outcome will be reported as an average score.

SECONDARY OUTCOMES:
Patient care | Data will be collected pre- and post-intervention for approximately 5 weeks total.
  Patient care delivered by subjects and their respective team during trauma resuscitations is video recorded and assessed using a patient care measure (behaviorally anchored rating scale). Final outcome will be reported as an average score.

OTHER OUTCOMES:
Survival to discharge | Data will be collected up to 4 months after admission
  defined as alive when left hospital or at 28 days, whichever comes first.
Total hospital length of stay | Data will be collected up to 4 months after admission
  calculated by subtracting the admission date from the discharge date. If a patient is admitted and discharged on the same date, the length of stay is calculated as one day.
Total intensive care length of stay | Data will be collected up to 4 months after admission
  calculated as the length of time spent in an intensive care unit in total hours divided by 24. Intensive care is defined as a ward of the hospital capable of providing mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemarie Fernandez, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No